CLINICAL TRIAL: NCT00873171
Title: Osteopathic Manipulation Therapy in the Treatment of Interstitial Cystitis
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: James P. Tierney DO., CAMC Medical Staff - with admitting privileges
Other Study IDs: 08-04-2046
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Interstitial Cystitis
Keywords: Osteopathic Manipulation
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1. OMT: This procedure consist of Sacral rocking is performed by placing the heel of the practitioner's hand over the sacrum and by using the palpatory skills of an osteopathic physician; rock the sacrum into a position with no restriction. Myofascial release will utilize various physical motions to place the patients lumbosacral region in a position of maximal comfort and tissue release.
- 2. Attention control OMT: The procedure consist of light pressure applied to certain painful areas of the body and back to decrease pain and help patient relax. The physician will look for areas of the body that hurt, lay his/her hands on the those places, and apply light pressure.
- 3. Standard of Care: This procedure consists of various conservative treatments that can help reduce stress. Those include dietary modifications, pharmaceuticals, bladder training, and neuromodulation. If these treatments are not successful, minimally invasive surgical procedures is performed.

SUMMARY:
As a safe and noninvasive method of treatment, the intent of the study is to show that Osteopathic manipulation therapy is a beneficial treatment for the aggravating bladder symptoms seen in all patients with interstitial cystitis.

DETAILED DESCRIPTION:
The management of interstitial cystitis is predominantly based on the reduction of the symptoms of frequency, urgency, and pain.In addition to Osteopathic manipulation Other conservative treatments frequently include dietary modification, pharmaceuticals, bladder training, neuromodulation, and stress reduction. The goal of Osteopathic manipulation is to relax the pelvic muscles used by the bladder and improve the flow of blood and lymph fluid to this region, which may result in easing pain and discomfort associated with cystitis.Some physicians have found that Osteopathic Manipulation works for some people as an alternative to surgery. A secondary objective will be to determine if the increased attention and power of touch are as effective as OMT in treating patients with interstitial cystitis based on the results of using attention control treatment in some patients.Thus, this is a pilot study comparing OMT to an attention control arm and standard of care arm of treatment.We will review palpatory visceromatic reflex changes as documented by tissue texture changes, asymmetry, restriction of motion and tenderness pre and post treatment.Physical examination including detailed musculoskeletal examination of the lumbosacral region will be performed pre and post and then compared the results.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for treatment is that the patient must exhibit symptoms of IC for at least one year and have a known diagnosis based on history and clinical findings including glomerulations of the bladder wall seen on cystoscopic examination.

Exclusion Criteria:

* Patients who are not eligible are those who have contraindications to OMT such as hypersensitivity to palpation, indurations or mass/tumor, adenopathy, cancer, or local infection

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample of 60 patients that have a confirmed diagnosis of Interstitial Cystitis as patients of Urological Surgical Associates and Charleston Area Medical Center (CAMC) based on current diagnostic recommendations. The patients will be selected based on their clinical history of interstitial cystitis.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Osteopathic Manipulation therapy over standard of care invasive procedures for the treatment of interstitial cystitis. | Within 2 weeks of treatment

SECONDARY OUTCOMES:
To determine if the increased attention and power of touch are as effective as OMT in treating patients with IC based on the results of using attention control treatment in some patients. | Within 2 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: James P Tierney, D.O., Principal Investigator — CAMC Medical Staff - with admitting privileges
Locations (1):
- James P. Tierney D.O., Charleston, West Virginia, United States